CLINICAL TRIAL: NCT00237458
Title: An Open-label Continuation Trial to Assess the Continued Efficacy and Safety of Ascending Doses of Lacosamide in Subjects With Chronic Refractory Neuropathic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP0647
Record Dates: First submitted 2005-10-11; First posted 2005-10-12 (Estimated); Results first posted 2012-05-15 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-07

CONDITIONS: Chronic Refractory Neuropathic Pain
MeSH Terms: interventions — Lacosamide; 2-(acetylamino)-3-methoxy-N-(phenylmethyl)-, (2R)-

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lacosamide (Experimental): Open-label active treatment
  Interventions: Drug: Lacosamide

INTERVENTIONS:
Drug: Lacosamide — Dosage: Lacosamide up to 400 mg/day;
  Dosage form: Film-coated tablets;
  Dosage Frequency and Duration: Two times per day; 9.5 years
  Other Names: SPM 927; Vimpat

SUMMARY:
This trial is the follow-on trial to a preceeding open-label trial which included patients with chronic refractory neuropathic pain. It is conducted at one site in the United Kingdom and the patient enrollment is completed. The patients had successfully completed the above mentioned trial and, in the investigator's opinion, would benefit from long-term administration of Lacosamide. After a 1-week run-in phase the patients were uptitrated to their optimal dose and then continued into the maintenance phase. Different pain qualities are assessed by a patient's diary.

ELIGIBILITY:
Inclusion Criteria:

* Subject is informed and given ample time and opportunity to think about her/his participation in this extension trial and has given her/his written informed consent
* Subject met all inclusion criteria defined in the SP611 trial with SPM927 at the time of enrollment into trial SP611
* Subject has successfully completed trial SP611 and, in the investigator's opinion, would benefit from long-term administration of SPM927
* Subject is willing and able to comply with all trial requirements, including the ability to complete trial questionnaires

Exclusion Criteria:

* Subject previously participated in this trial
* Subject has participated in another trial of an investigational drug within the last 3 months (excluding trial SP611) or is currently participating in another trial of an investigational drug
* Subject has had prior therapy with a Nonsteroidal Anti-inflammatory Drug (NSAID) or Anti-epileptic Drug (AED) within 28 days prior to the Eligibility Visit
* Subject has evidence or history of significant Cardiovascular Disease within 12 months prior to the Eligibility Visit
* Subject has laboratory values, which are outside the normal range and judged by the Investigator to be clinically significant
* Subject has abnormal Renal or Hepatic function
* Subject has a history of Malignancies with the exception of subjects with a documented disease-free interval of 5 years or more
* Subject has a history of chronic alcohol or drug abuse within the last 12 months
* Subject has any medical or psychiatric condition which, in the opinion of the Investigator, could jeopardize or compromise the subject's ability to participate in this continuation trial
* Subject with a known history of severe Anaphylactic Reaction and/or serious or life threatening Blood Dyscrasias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2001-05; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (1):
- Monheim, Germany

REFERENCES:
- [Result] McCleane G, Koch B, Rauschkolb C. Does SPM 927 have an analgesic effect in human neuropathic pain? An open label study. Neurosci Lett. 2003 Dec 4;352(2):117-20. doi: 10.1016/j.neulet.2003.08.036. PMID 14625037
- [Result] Shaibani A, Biton V, Rauck R, Koch B, Simpson J. Long-term oral lacosamide in painful diabetic neuropathy: a two-year open-label extension trial. Eur J Pain. 2009 May;13(5):458-63. doi: 10.1016/j.ejpain.2008.05.016. Epub 2008 Jul 10. PMID 18619874
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started in May 2001 with subjects from Germany. The primary completion date and study completion date occurred in March 2011.
Pre-assignment Details: One subject was discontinued on the study due to the Adverse Event of Vertigo. However, the Termination page of the Case Report Form reflected that the subject withdrew consent. Therefore, the Participant Flow will reflect 3 subjects did not complete the study, while the subjects withdrawing from Adverse Events will reflect 2.
Period: Overall Study
Arm/Group | Lacosamide
Started | 7
Completed | 4
Not Completed | 3
Not completed — Lack of Efficacy | 1
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lacosamide
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.4 (10.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Region of Enrollment [Number; unit: participants]
  Germany | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting At Least 1 Treatment-Emergent Adverse Event (TEAE) During The Treatment Period.
Time Frame: From Baseline Visit to Final Week of Treatment (approximately 10 years)
Population: Of the 7 subjects in the Safety Set (SS), 7 are included in this analysis.
Measure: Number; unit: participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 7
participants | 7

2. Primary Outcome: Number of Subjects Withdrawing From Study Due To A Treatment-Emergent Adverse Event (TEAE) During The Treatment Period.
Time Frame: From Baseline Visit to Final Week of Treatment (approximately 10 years)
Population: Of the 7 subjects in the Safety Set (SS), 7 are included in this analysis.
Measure: Number; unit: participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 7
participants | 2

3. Secondary Outcome: Within-Subject Change In Average Daily Pain Score During the Treatment Period.
Description: The Average Daily Pain Score is calculated using an 11-point Likert scale, ranging from 0 (no pain) to 10 (worst pain ever experienced).
Time Frame: From Baseline Visit to Final Week of Treatment (approximately 9 years)
Population: Of the 7 subjects in the Safety Set (SS), 7 are included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 7
units on a scale | -2.9 (3.38)

4. Secondary Outcome: Within-Subject Change In The Perception Of Each Of The Individual Cardinal Symptoms of Pain During The Treatment Period - Shooting.
Description: Each individual cardinal symptom of pain is calculated using an 11-point Likert scale, ranging from 0 (no pain) to 10 (worst possible pain).
Time Frame: From Baseline Visit to Final Week of Treatment (approximately 9 years)
Population: Of the 7 subjects in the Safety Set (SS), 7 are included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 7
units on a scale | -2.3 (4.27)

5. Secondary Outcome: Within-Subject Change In The Perception Of Each Of The Individual Cardinal Symptoms of Pain During The Treatment Period - Burning.
Description: as for outcome 4
Time Frame: From Baseline Visit to Final Week of Treatment (approximately 9 years)
Population: Of the 7 subjects in the Safety Set (SS), 7 are included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 7
units on a scale | 0.4 (2.15)

6. Secondary Outcome: Within-Subject Change In The Perception Of Each Of The Individual Cardinal Symptoms of Pain During The Treatment Period - Paraesthesiae.
Description: as for outcome 4
Time Frame: From Baseline Visit to Final Week of Treatment (approximately 9 years)
Population: Of the 7 subjects in the Safety Set (SS), 7 are included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 7
units on a scale | -2.1 (3.34)

7. Secondary Outcome: Within-Subject Change In The Perception Of Each Of The Individual Cardinal Symptoms of Pain During The Treatment Period - Numbness.
Description: as for outcome 4
Time Frame: From Baseline Visit to Final Week of Treatment (approximately 9 years)
Population: Of the 7 subjects in the Safety Set (SS), 7 are included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 7
units on a scale | -2.4 (3.78)

8. Secondary Outcome: Within-Subject Change In The Perception Of Each Of The Individual Cardinal Symptoms of Pain During The Treatment Period - Allodynia.
Description: Each individual cardinal symptom of pain is calculated using an 11-point Likert scale, ranging from 0 (no pain) to 10 (worst possible pain).
  Allodynia is defined as neuropathic pain caused by normally innocuous stimuli becoming painful.
Time Frame: From Baseline Visit to Final Week of Treatment (approximately 9 years)
Population: Of the 7 subjects in the Safety Set (SS), 7 are included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 7
units on a scale | 0.6 (2.37)

9. Secondary Outcome: Subject's Global Impression of Change In Pain During The Treatment Period.
Description: The Subject's Global Impression of Change is a self-evaluation by the subject of their overall change in relief of neuropathic pain since the beginning of the study rated on a 7-point scale ranging from:
  1. Much better
  2. Moderately better
  3. Mildly better
  4. No change
  5. Mildly worse
  6. Moderately worse
  7. Much worse
Time Frame: From Baseline Visit to Final Week of Treatment (approximately 9 years)
Population: Of the 7 subjects in the Safety Set (SS), 7 are included in this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 7
percentage of participants
  Better | 85.7
  No Change | 14.3
  Worse | 0

10. Secondary Outcome: Investigator's Global Impression of Change In Pain During The Treatment Period.
Description: The Investigator's Global Impression of Change is a physician's assessment of the patient's overall change in relief of neuropathic pain since the beginning of the study rated on a 7-point scale ranging from:
  1. Much better
  2. Moderately better
  3. Mildly better
  4. No change
  5. Mildly worse
  6. Moderately worse
  7. Much worse
Time Frame: From Baseline Visit to Final Week of Treatment (approximately 9 years)
Population: Of the 7 subjects in the Safety Set (SS), 7 are included in this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 7
percentage of participants
  Better | 85.7
  No Change | 14.3
  Worse | 0

11. Secondary Outcome: Percentage of Days With Concomitant Pain ("Rescue") Medications Taken During Baseline Phase.
Description: The percentage of days where rescue medication was taken is summarized by visit and by Treatment Phase (Baseline, Titration, and Titration + Treatment).
  The percentage of days of rescue medication use is defined as the number of days observed within the visit/study phase with rescue medication divided by the number of days in the visit/study phase times 100 for subjects who had taken the rescue medication.
  Summary statistics include mean and standard deviation.
Time Frame: Baseline Period (approximately 1 week)
Population: Of the 7 subjects in the Safety Set (SS), 4 are included in this analysis.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Lacosamide
Number analyzed (Participants) | 4
percentage of days | 100 (0.00)

12. Secondary Outcome: Percentage of Days With Concomitant Pain ("Rescue") Medications Taken During Titration Phase.
Description: as for outcome 11
Time Frame: Titration Period (approximately 6 weeks)
Population: Of the 7 subjects in the Safety Set (SS), 4 are included in this analysis.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Lacosamide
Number analyzed (Participants) | 4
percentage of days | 51.3 (36.98)

13. Secondary Outcome: Percentage of Days With Concomitant Pain ("Rescue") Medications Taken During Titration and Treatment Phases.
Description: as for outcome 11
Time Frame: From Titration Phase through Treatment Phase (approximately 9 years)
Population: Of the 7 subjects in the Safety Set (SS), 5 are included in this analysis.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Lacosamide
Number analyzed (Participants) | 5
percentage of days | 12.3 (7.91)

ADVERSE EVENTS:
Time Frame: The Time Frame for Adverse Event Reporting was the maximum exposure time of 9.5 years.
Arm/Group | Lacosamide
Serious Adverse Events (participants affected / at risk) | 4/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (N=7)
Chest Pain (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1)
Weight Decreased (Investigations) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Circulatory Collapse (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (N=7)
Sinus Bradycardia (Cardiac disorders) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Conjunctival Haemorrhage (Eye disorders) | 1 (1)
Iritis (Eye disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Enterocolitis Haemorrhagic (Gastrointestinal disorders) | 1 (1)
Peptic Ulcer (Gastrointestinal disorders) | 1 (1)
Stomach discomfort (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (3)
Influenza (Infections and infestations) | 2 (3)
Localised Infection (Infections and infestations) | 1 (1)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (1)
Mumps (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (5)
Pharyngitis (Infections and infestations) | 2 (4)
Sinusitis (Infections and infestations) | 1 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 3 (14)
Viral Infection (Infections and infestations) | 2 (3)
Foot Fracture (Injury, poisoning and procedural complications) | 1 (1)
Fractured Coccyx (Injury, poisoning and procedural complications) | 1 (1)
Joint Sprain (Injury, poisoning and procedural complications) | 1 (1)
Muscle Strain (Injury, poisoning and procedural complications) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 1 (1)
Basophil Count Increased (Investigations) | 1 (1)
Blood Phosphorus Increased (Investigations) | 1 (1)
Blood Sodium Decreased (Investigations) | 1 (1)
Electrocardiogram QT Corrected Interval Prolonged (Investigations) | 1 (2)
Electrocardiogram QT Prolonged (Investigations) | 1 (1)
Gamma-glutamyltransferase Increased (Investigations) | 1 (2)
Neutrophil Count Decreased (Investigations) | 3 (4)
Platelet Count Decreased (Investigations) | 2 (4)
Thyroxine Free Increased (Investigations) | 1 (1)
Diabetes Mellitus (Metabolism and nutrition disorders) | 2 (2)
Diabetes Mellitus Non-insulin-dependent (Metabolism and nutrition disorders) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 4 (5)
Headache (Nervous system disorders) | 2 (9)
Tension Headache (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Sleep disorder (Psychiatric disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that the results shall be published regardless of outcome.